CLINICAL TRIAL: NCT02323711
Title: A Randomized Controlled Trial of Dressing Versus Glue (2-Octyl Cyanoacrylate) for Coverage of the Skin Incision After Closure During Cesarean Delivery
Brief Title: Dressing Versus Glue (2-Octyl Cyanoacrylate) for Coverage of the Skin Incision After Closure During Cesarean Delivery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator Preference.
Sponsor: Danbury Hospital (Other)
Responsible Party: Principal Investigator, Matthew Kim, Section Chief, Maternal Fetal Medicine and Medical Director, Labor and Delivery, Department of Obstetrics, Gynecology, and Reproductive Services, Danbury Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: WCHN/IRB 13-56
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Pregnant Women; Cesarean Section

ARMS (2):
- Control (No Intervention): This group would be receiving the standard of care. The subject would receive the standard dressing applied by a member of the surgical team in the standard fashion as follows: The closed incision will be covered first with a primary dressing consisting of a nonadherent, composite dressing (Telfa), which is covered with a secondary dressing consisting of an Army Battle Dressing (ABD), before removal of the sterile surgical drapes. This dressing is then held in place with an adhesive fabric tape, currently Mefix tape, which is typically applied by the surgical scrub tech.
- 2-octyl cyanoacrylate (Experimental): This group would receive the experimental treatment. If allocated to coverage with glue, no dressing is placed. After closure of the incision with suture or staples, the incision is patted dry under sterile conditions. The incision is then covered longitudinally by a member of the surgical team with a thick layer of skin glue dispensed from 1 tube of surgical skin glue (2-octyl cyanoacrylate, currently using brand: Derma+Flex QS). The glue is then allowed to dry before the sterile surgical drapes are removed.
  Interventions: Device: 2-octyl cyanoacrylate

INTERVENTIONS:
Device: 2-octyl cyanoacrylate — If the subject is allocated to the experimental group, they would receive 2-octyl cyanoacrylate in place of a primary dressing consisting of their non-adherent composite dressing (Tefla) and a secondary dressing of Army Battle Dressing (ABD).
  Other Names: Derma+flex QS
  Arms: 2-octyl cyanoacrylate

SUMMARY:
This study is investigating the relative risks and benefits of using two common materials for coverage of the skin incision at cesarean delivery. We will perform the first prospective and the first randomized controlled trial examining the use of a standard postoperative dressing versus skin glue for coverage of the closed skin incision after cesarean delivery. The hypothesis is that using skin glue for coverage of the incision will be associated with decreased wound complications and increased patient satisfaction.

DETAILED DESCRIPTION:
Given the plethora of literature regarding technical aspects of performing cesarean delivery, and given the large number of procedures performed each year and available for prospective trials (approximately 700 cesarean deliveries per year at Danbury Hospital), only quality level I evidence is broadly considered influential in this area of research. Therefore we propose a RCT for incision coverage with dressing versus glue at cesarean delivery.

On admission to L&D for schedule cesarean section, or on admission to L&D for labor, patients will be asked to participate by a Trial Coordinator or the admitting Obstetrics and Gynecology resident physician. Patients admitted for labor will be asked to participate given the possibility that they may ultimately require cesarean delivery, and because using only patients admitted for scheduled cesarean delivery would eliminate urgent and emergent cesarean deliveries from the trial, and therefore decrease the generalizability of the trial results to general obstetrics practice.

When consented and the patient undergoes cesarean delivery, the patient's surgeon will decide if skin closure will be performed by placement of staples or suture. The circulating nurse in the OR will open one of a set of sequentially numbered, opaque sealed envelopes (SNOSE) to indicate the patient's allocation for coverage of the incision with a dressing or glue. The circulating nurse will then tell the surgeon to which group the patient has been allocated.

Before closure of the incision, care is taken to ensure hemostasis of the subcutaneous tissues and skin edges. If the subcutaneous tissues are > 2 cm thick, this tissue layer should be approximated before closure of the skin as is currently a level I evidence-based recommendation based on multiple RCTs and promoted by current clinical guidelines. Choice of suture material and needle for the running subcuticular closure, or use of staples for closure, are per the surgeon's preference.

If allocated to coverage with dressing, the standard dressing will be applied by a member of the surgical team in the standard fashion as follows: The closed incision will be covered first with a primary dressing consisting of a nonadherent, composite dressing (Telfa), which is covered with a secondary dressing consisting of an Army Battle Dressing (ABD), before removal of the sterile surgical drapes. This dressing is then held in place with an adhesive fabric tape, currently Mefix tape, which is typically applied by the surgical scrub tech.

If allocated to coverage with glue, no dressing is placed. After closure of the incision with suture or staples, the incision is patted dry under sterile conditions. The incision is then covered longitudinally by a member of the surgical team with a thick layer of skin glue dispensed from 1 tube of surgical skin glue (2-octyl cyanoacrylate, currently using brand: Derma+Flex QS). The glue is then allowed to dry before the sterile surgical drapes are removed.

Staples placed for incision closure are routinely removed on the day of discharge. Sutures placed for skin closure are absorbable and are therefore not removed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women admitted to Labor and Delivery for scheduled cesarean section, for labor, or for induction of labor
* Age >/= 18 years
* All gestational ages
* All numbers of gestations
* All fetal presentations
* All maternal and fetal medical or surgical comorbidities are included except as listed in the exclusion criteria

Exclusion Criteria:

* Patient is under 18 years of age.
* Intrauterine fetal death, excluded simply for social reasons concerning consenting the patient for the study during upsetting circumstances.
* Patient is NOT fluent in English, Spanish, or Portuguese.
* Urgent or emergent cesarean delivery for fetal distress that develops before the patient is approached for consent
* Patient incompetent to provide independent informed consent.
* Patient has a known allergy to Glue, Tape, Cyanoacrylate, and/or Formaldehyde.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Any Significant complications | 30 Days following cesarean delivery.
  the primary outcome of the study will be a composite outcome of any significant complications including wound separation, wound infection, symptomatic seroma or hematoma, or readmission for a wound complication within 30 days postoperatively. This data is gathered from the subject's medical record and from the Discharging Resident Questionnaire.

SECONDARY OUTCOMES:
Minor Complications and/or Patient Dissatisfaction | 30 Days following cesarean delivery
  Secondary outcomes will include problems with the periwound skin including blistering or skin tears, as well as pain or itching of the wound and periwound skin, narcotic use during the hospitalization, and overall patient satisfaction with the incision at the time of discharge. This data is gathered from the subject's medical record and the Patient Discharge Questionnaire, the Patient Follow-Up Questionnaire, and the Physician Follow-Up Questionnaire(if applicable).

REFERENCES:
- [Background] Romero P, Frongia G, Wingerter S, Holland-Cunz S. Prospective, randomized, controlled trial comparing a tissue adhesive (Dermabond) with adhesive strips (Steri-Strips) for the closure of laparoscopic trocar wounds in children. Eur J Pediatr Surg. 2011 May;21(3):159-62. doi: 10.1055/s-0030-1270458. Epub 2011 Jan 31. PMID 21283958
- [Background] Ong CC, Jacobsen AS, Joseph VT. Comparing wound closure using tissue glue versus subcuticular suture for pediatric surgical incisions: a prospective, randomised trial. Pediatr Surg Int. 2002 Sep;18(5-6):553-5. doi: 10.1007/s00383-002-0728-0. Epub 2002 Jun 14. PMID 12415411
- [Background] Cho J, Harrop J, Veznadaroglu E, Andrews DW. Concomitant use of computer image guidance, linear or sigmoid incisions after minimal shave, and liquid wound dressing with 2-octyl cyanoacrylate for tumor craniotomy or craniectomy: analysis of 225 consecutive surgical cases with antecedent historical control at one institution. Neurosurgery. 2003 Apr;52(4):832-40; discussion 840-1. doi: 10.1227/01.neu.0000054219.35102.b4. PMID 12657178
- [Background] Rajimwale A, Golden BK, Oottomasathien S, Krishnamurthy M, Ullrich NO, Koyle MA. Octyl-2-cyanoacrylate as a routine dressing after open pediatric urological procedures. J Urol. 2004 Jun;171(6 Pt 1):2407-8. doi: 10.1097/01.ju.0000125221.50141.33. PMID 15126862
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683
- [Background] Singer AJ, Hollander JE, Valentine SM, Turque TW, McCuskey CF, Quinn JV. Prospective, randomized, controlled trial of tissue adhesive (2-octylcyanoacrylate) vs standard wound closure techniques for laceration repair. Stony Brook Octylcyanoacrylate Study Group. Acad Emerg Med. 1998 Feb;5(2):94-9. doi: 10.1111/j.1553-2712.1998.tb02590.x. PMID 9492126
- [Background] Siddiqui DS, Lacuna EM, Chen HY, Chauhan SP. Skin closure of pfannenstiel incision with dermabond, staples, or suture during cesarean delivery: experience of a single attending. Am J Perinatol. 2013 Mar;30(3):219-24. doi: 10.1055/s-0032-1323583. Epub 2012 Aug 8. PMID 22875661
- [Background] Aabakke AJM, Krebs L, Pipper CB, Secher NJ. Subcuticular suture compared with staples for skin closure after cesarean delivery: a randomized controlled trial. Obstet Gynecol. 2013 Oct;122(4):878-884. doi: 10.1097/AOG.0b013e3182a5f0c3. PMID 24084548